CLINICAL TRIAL: NCT05309720
Title: Dermal Substitution in Paediatric Burns: A Prospective Case Series
Brief Title: Dermal Substitution in Pediatric Burns
Acronym: GlyPeB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-13625
Record Dates: First submitted 2022-03-15; First posted 2022-04-04 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-11

CONDITIONS: Burns; Burn Scar
Keywords: Burns; Scar quality; Pediatric
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: prospective case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glyaderm (Experimental)
  Interventions: Procedure: Glyaderm

INTERVENTIONS:
Procedure: Glyaderm — All included patients will undergo full thickness removal of the burned skin or adequate debridement of all necrotic tissue. Next, the dermal substitute Glyaderm followed by a split thickness skin graft will be transplanted on the wound.

SUMMARY:
The standard treatment of deep dermal to full thickness burns is surgical removal of the burn followed by skin transplantation. Dermal substitutes are increasingly used in the treatment of deep burns to replace lost dermis. Preservation of the collagen and elastin in the acellular human dermal substitute Glyaderm provides a more elastic scar. It is unknown what the effect of Glyaderm on scar quality is in a solely paediatric population.

The objective of this case series is to investigate scar maturation and scar quality when applying Glyaderm in deep dermal to full thickness burns in a pediatric population aged ≤15 years old.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤15 years old
2. Burn wounds requiring skin grafting
3. Written informed consent provided by

   1. The participant's parent(s)/guardian (<12 years of age)
   2. The participant's parent(s)/guardian and the participant itself (12-15 years old)

Exclusion Criteria:

1. Burn wound of ≤30 cm2
2. Infected burn wounds: clinical symptoms in combination with positive wound swabs
3. Patients/parents with insufficient knowledge of the Dutch or English language, since they would not be able to complete the POSAS questionnaire.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Scar quality (clinician) | 12 months
  Scar quality measured using the Patient and Observer Scar Assessment Scale (POSAS) Observer Scale, which rates the scar from 1 (=like normal skin) to 10 (=worst scar imaginable).

SECONDARY OUTCOMES:
Clinical assessment of the graft take | 5-7 days after STSG application
  Take of the split thickness skin graft (STSG) in percentages. The take is defined as STSG that appears vital and is adherent to the wound bed.
Wound epithelialization | 5-7 days after STSG application
  Wound epithelialization is the percentage of the graft with a vital skin graft and healed graft interstices.
Wound healing time | determined in the first several days to weeks after STSG application
  >95% epithelialization of the wound area is considered as healed
Donor site healing time | determined in the first several days to weeks after STSG application
  >95% epithelialisation of the donor site wound surface area is considered as healed
Scar surface area | day of surgery (day 0) and 3, 6 and 12 months post-surgery
  The scar surface area is calculated using the surgery wound as reference area
Scar quality (participant) | 3, 6 and 12 months post-surgery
  Scar quality measured using the Patient and Observer Scar Assessment Scale (POSAS) Patient Scale, rating the scar from 1 (=like normal skin) to 10 (=worst scar imaginable).
Occurrence of scar contractures | Up to 12 months post-surgery
  Scar contractures often occur in children with deep dermal and full thickness burn wounds.
Occurrence of scar hypertrophy | Up to 12 months post-surgery
  Scar hypertrophy often occurs in children with deep dermal and full thickness burn wounds.
Range of motion of affected joints | 3, 6 and 12 months post-surgery
  When joints are affected due to the burn wound, the range of motion of the affected joint(s) will be monitored during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Vehmeijer-Heeman, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided